CLINICAL TRIAL: NCT06668116
Title: The Impact of Local Anesthetic Dilution on the Possibility of Blinding Studies Involving Peripheral Nerve Blocks. A Randomized, Prospective, Monocentric Study on Volunteers
Brief Title: The Impact of Local Anesthetic Dilution on Possible Blinding for Nerve Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2024-01431
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Healthy
Keywords: Peripheral nerve blocks; Placebo-controlled studies; Blinding in clinical trials

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine-Placebo Arm (Other): Participants will first receive a nerve block with ropivacaine, starting at 0.1% concentration and adjusted according to Dixon's up-and-down method as described in the intervention section. Pain sensitivity and presence of sensory or motor block will be assessed 60 minutes post-injection using a Numerical Rating Scale (NRS). After a washout period, participants will cross over to receive a placebo (saline) injection, followed by the same assessments.
  Interventions: Drug: Ropivacaine 0,1%; Other: NaCl (placebo)
- Placebo-Ropivacaine Arm (Other): Participants will first receive a placebo (saline) nerve block injection. Pain sensitivity and any reported sensory or motor changes will be assessed 60 minutes post-injection using a Numerical Rating Scale (NRS). After a washout period, participants will cross over to receive the ropivacaine injection, with concentration determined by Dixon's up-and-down method as described in the intervention section, followed by the same assessments.
  Interventions: Drug: Ropivacaine 0,1%; Other: NaCl (placebo)

INTERVENTIONS:
Drug: Ropivacaine 0,1% — The study uses ropivacaine for nerve blocks, starting at 0.1% concentration and capped at 0.5% for safety. Concentration adjustments are made based on each participant's response 60 minutes post-injection:
  * Increase by 0.025% if pain reduction is <50%
  * Increase by 0.025% if reduction is 50-75% without sensory/motor block
  * Decrease by 0.025% if reduction is 50-75% with sensory/motor block
  * Decrease by 0.025% if reduction is >75%. Pain is assessed using a Numerical Rating Scale. The study employs Dixon's up-and-down method for five cycles to determine the optimal concentration for effective pain relief without significant numbness or weakness.
Other: NaCl (placebo) — 0.9 % NaCl solution (saline) injection

SUMMARY:
This study aims to determine the appropriate dosage of a placebo anesthetic to enable future placebo-controlled studies that can more accurately examine the effects of nerve blocks. The main challenge in conducting such studies is the difficulty in blinding participants and researchers due to the noticeable effects of nerve blocks, such as numbness and motor impairments.

The goal is to find a placebo solution that can:

* Mimic the sensations of a real nerve block
* Not provide actual pain relief
* Allow for effective blinding in future studies

By developing an appropriate placebo, researchers hope to:

* Enable more rigorous investigations into the efficacy of nerve blocks for pain management
* Conduct comprehensive placebo-controlled studies, which are currently lacking in the field
* Overcome the obstacle of ensuring successful blinding in nerve block research This study is focused to establish a methodology for creating a convincing placebo that can be used in future research to more accurately assess the true effects of nerve blocks in pain medicine.

DETAILED DESCRIPTION:
Nerve blocks are medical procedures commonly used in pain management for three main purposes: diagnosis, prognosis, and treatment. For diagnostic nerve blocks, the goal is to identify the source of pain. The underlying idea is straightforward: if numbing a specific nerve stops the pain, that nerve is likely the source of the problem. Conversely, if the pain persists after the nerve is numbed, it suggests that the issue lies elsewhere.

Prognostic nerve blocks serve a different function; they are used to test whether a future treatment might be successful. If a temporary nerve block alleviates pain, it indicates that a more permanent treatment targeting that nerve could be effective. Therapeutic nerve blocks aim to provide long-lasting pain relief, helping patients engage in physical therapy or acting as a treatment on their own.

Despite their widespread use, there is insufficient solid scientific evidence to fully support the effectiveness of nerve blocks. Most studies conducted so far rely on observational data rather than controlled experiments. This lack of robust evidence raises concerns because diagnostic and prognostic blocks may lead to incorrect diagnoses or ineffective treatments. Additionally, therapeutic blocks can be invasive and costly, yet their effectiveness is not always guaranteed.

One significant challenge in researching nerve blocks is the difficulty of conducting placebo-controlled studies. For these studies to be valid, researchers need to ensure that neither the patients nor the assessors know who received the actual treatment and who received a placebo. However, this is complicated by the fact that nerve blocks often cause noticeable numbness or weakness, making it easy to identify who received the real treatment.

Researchers are exploring the possibility of using very low doses of anesthetic that might provide pain relief without causing noticeable numbness or weakness. If successful, this approach could allow for proper "blinded" studies where neither patients nor researchers can tell who received the actual treatment.

In summary, while nerve blocks play an important role in pain medicine, more research is needed to confirm their effectiveness. Finding ways to conduct proper placebo-controlled studies is crucial for ensuring that these treatments truly benefit patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA I - II, both sexes
* ≥ 18 years old
* < 65 years old
* Written informed consent as documented by signature

Exclusion Criteria:

* Known allergy or hypersensitivity to a ropivacaine, amide local anesthetics or ultrasound gel
* Any history of chronic or acute pain at the moment of enrollment into the study
* Treatment with any substance having a relation to pain or pain modulation (antidepressants, opioids, benzodiazepines, anticonvulsants)
* Intake of any analgesic 48 hours prior to the conduction of any of the study stages
* Severe coagulopathy
* History of cardiovascular disease
* History of alcohol abuse or the intake of psychotropic drugs
* Pregnancy, ruled out by history
* Infection at the injection site or a systemic infection
* Fever of unknown origin
* Motor or sensory abnormalities in the arm
* Previous enrollment into the current study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2024-12-11 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Heat pain sensitivity | Heat pain sensitivity will be determined before (baseline), and every 5 minutes up to 60 minutes after injection.
  Participants will rate their pain in response to heat stimulation using the Numerical Rating Scale (NRS). On this scale, 0 represents no pain at all, while 100 represents the worst pain imaginable.
Self-report of sensory block | Self-report of sensory block will be assessed 30 and 60 minutes after injections.
  Participants will be asked to self-report any sensory changes by responding to the question: "Do you feel any numbness in the forearm or hand on the side where the injection was given?" They will be required to answer either "yes" or "no" to this question.
Self-report of motor block | Self-report of motor block will be assessed 30 and 60 minutes after injections.
  Participants will be asked to self-report any motor changes by responding to the question: "Do you feel any reduction of strength of your hand on the injection side?" They will be required to answer either "yes" or "no" to this question.

SECONDARY OUTCOMES:
Evaluation of the C-fiber block | Measurement will be done at baseline, 30 and 60 minutes after injection.
  C-fibers will be evaluated by measuring electrodermal activity, specifically continuous skin conductance level and phasic heat-induced sympathetic skin response (SSR). These measurements will be taken in the innervation area of the ulnar nerve, specifically at the digitus minimus of the non-dominant hand, using Ag/AgCl electrodes filled with a skin conductance electrode paste. Phasic sympathetic skin response will be induced by applying five heat stimuli ranging from 42 to 52°C to the contralateral volar forearm. Electrodermal activity will be recorded using LabChart data acquisition software and PowerLab hardware. Participants will be instructed to relax and lie quietly in a supine position, with the ambient temperature maintained between 22-24°C. Continuous skin conductance level measurements will begin at baseline and continue throughout the injection until the signal disappears, at which point the time to signal disappearance will be recorded.
Evaluation of the A-delta fiber block | Measurement will be done at baseline, 30 and 60 minutes after the injection.
  To evaluate the block of the A-delta fibers of the ulnar nerve, five heat stimuli will be applied within the innervation area of the ulnar nerve (same as for heat pain sensitivity described above) and the phasic heat-induced sympathetic skin response from the contralateral palm will be recorded.
Evaluation of the A-beta fiber block | Measurement will be done at baseline, 30 and 60 minutes after the injection.
  The function of A-beta fibers will be tested using ulnar somatosensory evoked potentials (SSEPs). Measurements will be conducted while participants are in a supine position, following the guidelines of the German Society for Clinical Electrophysiology and Medical Imaging. Electrical stimulation of the ulnar nerve at the hypothenar eminence of the non-dominant hand will be applied using the Dantec Keypoint® 4 System through self-adhesive surface electrodes. The stimulation intensity will be set at four times the electrical perception threshold, with a frequency of 3.1 Hz and a pulse width of 0.2 milliseconds. SSEPs will be recorded by the same system through needle electrodes placed over Fz (as reference) and C3'/C4', according to the international 10-20 EEG electrode positioning system. Signals will be recorded at a frequency of 12 kHz and band-pass filtered between 500 Hz and 1 kHz, with N20 latencies and amplitudes of the N20/P25 complex manually detected.
Evaluation of the A-alpha fiber block (motor block) | Measurement will be done at baseline, 30 and 60 minutes after the injection.
  Motor block of the ulnar nerve will be evaluated using motor nerve conduction studies performed according to clinical standards (see Neurophysiology Manual used within EMSCI, ww.emsci.org). Compound motor action potentials (cMAP) of the abductor digitimi minimi (ADM) muscles will be recorded with surface electrodes (Ambu® BlueSensor NF, Ballerup, Denmark) with the active electrode placed over the motor point of the ADM and the reference electrode at the base of the fourth digit. cMAPs will be recorded with a sampling rate of 2000Hz and a bandpass filter of 5Hz-10kHz using the Dantec Keypoint® 4 System (Natus Medical Incorporated, San Carlos, CA, USA). The ulnar nerve at the proximal arm will be stimulated with a stimulation intensity of supramaximal level (1-100mA) and a constant current rectangular stimulation pulse of 0.2ms pulse width
Offset analgesia | Measurement will be done at 60 minutes after the injection.
  The evaluation of offset analgesia will follow published paradigms16,17 where a disproportionally large reduction in perceived pain following a slight decrease in painful stimulus intensity will be recorded. We will use a surface contact heat stimulator (PATHWAY Pain & Sensory Evaluation System, Medoc, Ramat Yishai, Israel) with the ATS thermode (30x30mm). We will attach the thermode to hypothenar eminence and ramped up from 35° to 47°C, then held for 5s at 47°C, increased to 48°C for 5s and decreased again to 47°C for 20s. We will use a computerized visual analogue scale (CoVAS, Medoc, Ramat Yishai, Israel) to get concomitant pain ratings during the paradigm.

OTHER OUTCOMES:
Evaluating blinding of the participants_part1 | Measurement will be done 60 minutes after the injection.
  To evaluate the effectiveness of blinding, participants will be asked which solution they believe they received, with response options of either "local anesthetic" or "saline."
Evaluating blinding of the participants_part2 | Measurement will be done 60 minutes after the injection.
  To assess the effectiveness of blinding, participants will be asked to express their level of certainty in response to the question, "Which solution do you believe you received?" Possible responses will include "completely certain," "partly certain," or "uncertain."

CONTACTS AND LOCATIONS:
Overall Officials: Hagen Bomberg, Medical Doctor, Principal Investigator — Deputy Head of Anesthesiology
Locations (1):
- Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Curatolo M, Petersen-Felix S, Arendt-Nielsen L. Sensory assessment of regional analgesia in humans: a review of methods and applications. Anesthesiology. 2000 Dec;93(6):1517-30. doi: 10.1097/00000542-200012000-00025. No abstract available. PMID 11149448
- [Background] Sveticic G, Gentilini A, Eichenberger U, Zanderigo E, Sartori V, Luginbuhl M, Curatolo M. Combinations of bupivacaine, fentanyl, and clonidine for lumbar epidural postoperative analgesia: a novel optimization procedure. Anesthesiology. 2004 Dec;101(6):1381-93. doi: 10.1097/00000542-200412000-00019. PMID 15564946
- [Background] Curatolo M, Kaufmann R, Petersen-Felix S, Arendt-Nielsen L, Scaramozzino P, Zbinden AM. Block of pinprick and cold sensation poorly correlate with relief of postoperative pain during epidural analgesia. Clin J Pain. 1999 Mar;15(1):6-12. doi: 10.1097/00002508-199903000-00003. PMID 10206562
- [Background] Vadhanan P, Tripaty DK, Adinarayanan S. Physiological and pharmacologic aspects of peripheral nerve blocks. J Anaesthesiol Clin Pharmacol. 2015 Jul-Sep;31(3):384-93. doi: 10.4103/0970-9185.161679. PMID 26330722
- [Background] Curatolo M, Schnider TW, Petersen-Felix S, Weiss S, Signer C, Scaramozzino P, Zbinden AM. A direct search procedure to optimize combinations of epidural bupivacaine, fentanyl, and clonidine for postoperative analgesia. Anesthesiology. 2000 Feb;92(2):325-37. doi: 10.1097/00000542-200002000-00012. PMID 10691217
- [Background] Inan LE, Inan N, Karadas O, Gul HL, Erdemoglu AK, Turkel Y, Akyol A. Greater occipital nerve blockade for the treatment of chronic migraine: a randomized, multicenter, double-blind, and placebo-controlled study. Acta Neurol Scand. 2015 Oct;132(4):270-7. doi: 10.1111/ane.12393. Epub 2015 Mar 13. PMID 25765043
- [Background] Dahan TH, Fortin L, Pelletier M, Petit M, Vadeboncoeur R, Suissa S. Double blind randomized clinical trial examining the efficacy of bupivacaine suprascapular nerve blocks in frozen shoulder. J Rheumatol. 2000 Jun;27(6):1464-9. PMID 10852272
- [Background] Adey-Wakeling Z, Crotty M, Shanahan EM. Suprascapular nerve block for shoulder pain in the first year after stroke: a randomized controlled trial. Stroke. 2013 Nov;44(11):3136-41. doi: 10.1161/STROKEAHA.113.002471. Epub 2013 Aug 22. PMID 23970790
- [Background] Lord SM, Barnsley L, Bogduk N. The utility of comparative local anesthetic blocks versus placebo-controlled blocks for the diagnosis of cervical zygapophysial joint pain. Clin J Pain. 1995 Sep;11(3):208-13. doi: 10.1097/00002508-199509000-00008. PMID 8535040
- [Background] Engel A, MacVicar J, Bogduk N. A philosophical foundation for diagnostic blocks, with criteria for their validation. Pain Med. 2014 Jun;15(6):998-1006. doi: 10.1111/pme.12436. Epub 2014 Apr 9. PMID 24716821